CLINICAL TRIAL: NCT00262262
Title: The Effect of Levetiracetam on the Postmastectomy Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIIS; PubliRC CNS 085 TA 1007 LEV
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Levetiracetam; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam (drug) — The starting dose of levetiracetam was 500 mg/day and the dose was increased with 500 mg every other day to 6 tablets of 500 mg (Keppra, UCB, Belgium), divided into two doses daily corresponding to 3000 mg/day. The dose was kept at this level throughout the remaining treatment period - 4 weeks total. Six placebo tablets with identical appearance were dosed similarly to levetiracetam in the placebo phase.
  Other Names: Keppra, Levetiracetam

SUMMARY:
The aim of this study is determine whether or not the antiepileptic drug Levetiracetam is an effective treatment of the postmastectomy pain syndrome.

DETAILED DESCRIPTION:
This study is a randomised, placebocontrolled, doubleblind study on the effect of the antiepileptic drug, levetiracetam, in patients suffering from PMPS. The treatment periods are 1 month each and the periods are separated by a 1-week washout period. The daily dose of levetiracetam is increased over a 2-week period to 3.000 mg/day. The primary effect variable is pain relief by the use of numeric rating scale. Secondary parameters are daily registration of pain performed by the patients during the treatment periods and the amount of escape medicine used (paracetamol and tramadol). Sensory testing is performed at baseline and after each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms characteristic for postmastectomy pain syndrome with a duration of more than 3 months and at least 6 months after the operation.
* Neuropathic pain diagnose confirmed by abnormities in the neurological investigation and/or psychophysical sensory testing
* Average (1 week) pain score minimum 4 on a 11 points numerical rating scale for total pain.
* Pain present minimum 4 out of 7 days.
* Fertile women must use anticonception.

Exclusion Criteria:

* Verified og suspected other reason than mastectomy/lumpectomy for the pain.
* Known allergic effects to levetiracetam.
* Known sideeffects to treatment with levetiracetam.
* Pregnancy or breast-feeding.
* Severe disease (terminal cancer, heart failure, kidney insufficiency, severe respiratory problems)
* Compliance problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Pain relief | After 1 month treatment

SECONDARY OUTCOMES:
Pain intensity measured daily on numeric rating scales | During treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Ole J Vilholm, MD, Study Director — Odense University Hospital; Søren H Sindrup, Professor MD, Principal Investigator — Odense University Hospital; Søren Cold, MD, Study Chair — Department of oncology, Odense University Hospital, Denmark; Lars Rasmussen, MD, Study Chair — Department of surgery, Odense University Hospital, Denmark
Locations (1):
- Department of neurology, Odense Universityhospital, Odense, Fyn, Denmark